CLINICAL TRIAL: NCT04108754
Title: Small-vessel Disease Burden and Early Risk of Stroke After Transient Ischemic Attack
Acronym: TIA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: TIA
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Diagnosis of TIA; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosis of AIT: Patients in the neurovascular unit of the Neurological Hospital of Lyon between 01/01/2016 and 30/12/2017 with a probable diagnosis of AIT and having an MRI within 7 days of TIA.
  Interventions: Other: microangiopathic burden

INTERVENTIONS:
Other: microangiopathic burden — to determine the value of the global microangiopathic burden on the prediction of early stroke risk in a homogeneous cohort of TIA.

SUMMARY:
Predicting the risk of stroke remains a challenge in the management of transient ischemic attack (TIA). In addition to clinical variables, morphological features such as the presence of a diffusion weighted sequence (DWI) lesion and carotid stenosis of at least 50% improve risk stratification and are considered in the literature. score ABCD3-I1. Several studies have shown that brain microhemorrhages are associated with the risk of early stroke in patients with TIA. Data on white matter hypersignals on the T2-weighted sequence or FLAIR (FLuid Attenuated Inversion Recovery) are more conflicting. The global microangiopathic load, including the gaps, the hypersignals of the white matter, the perivascular spaces visible on MRI in the basal ganglia, especially when they are very numerous (> 20) and the gaps, have recently been described as being associated with stroke risk within 2 to 3 years of TIA or ischemic stroke. To date, the predictive value of global microangiopathic burden on early stroke risk in the course of TIA is not known.

ELIGIBILITY:
Inclusion Criteria:

* Patients with probable TIA with Regression of symptoms within 24 hours (unilateral motor or sensory disorders affecting the face and / or limbs , language disorder, blindness of an eye or amputation of a visual field)
* Patients with possible AIT with 2 of these symptoms associated: fear of heights, diplopia, dysarthria, disorders of swallowing, loss of balance, isolated sensory symptoms affecting only part of a limb or hemiface.
* Patient who have had a brain MRI.
* Patient over 18 year-old.
* Patient who give their non opposition to participate at the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the neurovascular unit of the Neurological Hospital of Lyon between 01/01/2016 and 30/12/2017 with a probable diagnosis of TIA and having an MRI within 7 days of the TIA.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
stroke recurrence within 90 days, | 90 days
  The stroke recurrence within 90 days is determined via a clinical consultation or telephone call to the patient with a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert NIGHOGHOSSIAN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No